CLINICAL TRIAL: NCT07207876
Title: Phase IV Study of the Pharmacokinetics and Safety of Ceftriaxone and Benzathine Penicillin G During Pregnancy
Brief Title: Study of Ceftriaxone and Benzathine Penicillin G During Pregnancy
Status: Recruiting | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT 2044; UM1AI068632 (NIH); UM1AI068616 (NIH); UM1AI106716 (NIH); HHSN275201800001I (Other: Eunice Kennedy Shriver National Institute of Child Health and Human Development)
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy
Keywords: Cefriaxone; Syphilis; Pregnancy; Benzathine Penicillin G
MeSH Terms: conditions — Syphilis | interventions — Ceftriaxone; Penicillin G

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Active comparator: Arm 1A: IV ceftriaxone: Intravenous ceftriaxone
  Interventions: Drug: Ceftriaxon
- Active Comparator: Arm 1B: IM ceftriaxone: Intramuscular ceftriaxone
  Interventions: Drug: Ceftriaxon
- Active Comparator: Arm 2: IM benzathine penicillin G: Intramuscular benzathine penicillin G
  Interventions: Drug: Benzathine penicillin G

INTERVENTIONS:
Drug: Ceftriaxon — Ceftriaxone will not be provided as part of the study. Pregnant participants will receive these drugs as prescribed outside the study by their non-study clinical care provider
  Groups: Active Comparator: Arm 1B: IM ceftriaxone; Active comparator: Arm 1A: IV ceftriaxone
Drug: Benzathine penicillin G — Benzathine penicillin G will not be provided as part of the study. Pregnant participants will receive these drugs as prescribed outside the study by their non-study clinical care provider
  Groups: Active Comparator: Arm 2: IM benzathine penicillin G

SUMMARY:
IMPAACT 2044 is a study to characterize the pharmacokinetics (PK) and safety of ceftriaxone and benzathine penicillin G during pregnancy. Up to 78 pregnant women receiving (1) ceftriaxone for indications other than syphilis or (2) benzathine penicillin G for treatment of syphilis from non-study clinical care providers will be enrolled at study sites located in the United States. Approximately 22 infants of pregnant participants receiving benzathine penicillin G will also be enrolled.

DETAILED DESCRIPTION:
IMPAACT 2044 is a Phase IV, multi-site, open-label, non-randomized, opportunistic study to characterize the pharmacokinetics (PK) and safety of ceftriaxone and benzathine penicillin G during pregnancy.

The study includes two arms, with Arm 1 subdivided by route of administration:

Arm 1A: Intravenous (IV) ceftriaxone Arm 1B: Intramuscular (IM) ceftriaxone Arm 2: IM benzathine penicillin G

ELIGIBILITY:
Inclusion Criteria:

* Is of legal age or circumstance to provide independent informed consent as determined by site standard operating procedures (SOPs) and consistent with Institutional Review Board (IRB) policies and procedures and is willing and able to provide written informed consent for her own and, if applicable (Arm 2), her infant's study participation
* At screening, has a viable singleton intrauterine pregnancy of any gestational age confirmed by fetal ultrasound, as determined by the site investigator based on medical records, with trimester documented based on the best available obstetric estimate
* At screening, is receiving or expected to receive one of the following drugs under study as prescribed by a clinical care provider and documented in medical records:

  * Ceftriaxone: IV or IM administration for an indication other than syphilis
  * Benzathine penicillin G: IM administration for treatment of syphilis
* At entry, expects to remain in the geographic area of the study site during pregnancy and at least 30 days postpartum

Exclusion Criteria:

* Previously enrolled in this study
* Requires desensitization to ceftriaxone or benzathine penicillin G as determined by the site investigator based on pregnant participant report and available medical records
* Has any of the following as determined by the site investigator based on pregnant participant report and available medical records:

  * Current indication for hemodialysis
  * Current indication for intensive care unit hospitalization
  * Creatinine (Cr) ≥ 3.5 x upper limit of normal (ULN) at any time during the current pregnancy and/or chronic kidney disease Stage 5
* Receipt of any of the following prohibited medications within seven days prior to entry as determined by the site investigator based on pregnant participant report and available medical records:

  * Probenecid
  * Penicillin
* Arm 1A: any penicillin
* Arm 1B: any penicillin
* Arm 2: penicillin other than benzathine penicillin G

  * Benzapril
  * Chlorpropamide
  * Diflunisal
  * Irbesartan
  * Ketoprofen
  * Ketorolac tromethamine
  * Meclofenamic acid
  * Mefenamic acid
  * Oxaprozin
  * Parecoxib
  * Penciclovir
  * Pioglitazone
  * Telmisartan
  * Valsartan
* Receipt of any investigational agent within seven days prior to entry as determined by the site investigator based on pregnant participant report and available medical records
* Has any documented or suspected clinically significant condition that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women receiving or expecting to receive ceftriaxone for indications other than syphilis or benzathine penicillin G for treatment of syphilis during pregnancy in the United States (US). The infants of pregnant participants receiving benzathine penicillin G will also be enrolled.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Geometric mean area under the curve (AUC) during the dosing interval (AUC0-tau) in the first trimester trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean terminal elimination half-life (t1/2) in the first trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean trough concentration (Ctrough) in the first trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean AUC0-tau in the second trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean t1/2 in the second trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean Ctrough in the second trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean AUC0-tau in the third trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean t1/2 in the third trimester | First on-study dose through 24 hours
  Arm 1A
Geometric mean Ctrough in the third trimester | First on-study dose through 24 hours
  Arm 1A
Median maximum plasma concentration during the dose interval (Cmax) in the first trimester | First on-study dose through up to 24 hours
  Arm 1B
Median time to Cmax (Tmax) in the first trimester | First on-study dose through up to 24 hours
  Arm 1B
Median Cmax in the second trimester | First on-study dose through up to 24 hours
  Arm 1B
Median Tmax in the second trimester | First on-study dose through up to 24 hours
  Arm 1B
Median Cmax in the third trimester | First on-study dose through up to 24 hours
  Arm 1B
Median Tmax in the third trimester | First on-study dose through up to 24 hours
  Arm 1B
Geometric mean AUC at 7 days (AUC 0-7d) in the first trimester | First on-study dose through 7 days
  Arm 2
Geometric mean AUC at 14 days (AUC0-14d) in the first trimester | First on-study dose through 14 days
  Arm 2
Geometric mean plasma concentration at 2 hours (C2h) in the first trimester | 2 hours post-first on-study dose
  Arm 2
Geometric mean plasma concentration at 24 hours (C24h) in the first trimester | 24 hours post-first on-study dose
  Arm 2
Geometric mean plasma concentration at 4 days (C4d) in the first trimester | 4 days post-first on-study dose
  Arm 2
Geometric mean plasma concentration at 7 days (C7d) in the first trimester | 7 days post-first on-study dose
  Arm 2
Geometric mean plasma concentration at 14 days (C14d) in the first trimester | 14 days post-first on-study dose
  Arm 2
Geometric mean AUC0-7d in the second trimester | First on-study dose through 7 days
  Arm 2
Geometric mean AUC0-14d in the second trimester | First on-study dose through 14 days
  Arm 2
Geometric mean C2h in the second trimester | 2 hours post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C24h in the second trimester | 24 hours post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C4d in the second trimester | 4 days post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C7d in the second trimester | 7 days post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C14d in the second trimester | 14 days post-first on-study dose
  Arm 2 (as defined above)
Geometric mean AUC0-7d in the third trimester | First on-study dose through 7 days
  Arm 2
Geometric mean AUC0-14d in the third trimester | First on-study dose through 14 days
  Arm 2
Geometric mean C2h in the third trimester | 2 hours post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C24h in the third trimester | 24 hours post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C4d in the third trimester | 4 days post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C7d in the third trimester | 7 days post-first on-study dose
  Arm 2 (as defined above)
Geometric mean C14d in the third trimester | 14 days post-first on-study dose
  Arm 2 (as defined above)

SECONDARY OUTCOMES:
Proportion of participants with a maternal serious adverse event (SAE) | First on-study dose through 7 days
  Arm 1A and Arm 1B
Proportion of participants with a maternal SAE assessed as related to drug under study | First on-study dose through 7 days
  Arm 1A and Arm 1B
Proportion of participants with a maternal SAE | First on-study dose through up to 28 days
  Arm 2
Proportion of participants with a maternal SAE assessed as related to drug under study | First on-study dose through up to 28 days
  Arm 2
Proportion of participants with a spontaneous abortion or miscarriage (<20 weeks gestation) | At pregnancy outcome/delivery/birth
  Arm 1A, Arm1B, and Arm 2
Proportion of participants with a stillbirth (≥20 weeks gestation) | At pregnancy outcome/delivery/birth
  Arm 1A, Arm1B, and Arm 2
Proportion of participants with an infant small for gestational age (SGA; weight <10th percentile for gestational age, adjusted for sex) | At pregnancy outcome/delivery/birth
  Arm 1A, Arm1B, and Arm 2
Proportion of participants with a preterm birth (<37 weeks gestation) | At pregnancy outcome/delivery/birth
  Arm 1A, Arm1B, and Arm 2
Proportion of participants with an infant congenital anomaly consistent with the definition of defect provided by Metropolitan Atlanta Congenital Defects Program (MACDP) | At pregnancy outcome/delivery/birth
  Arm 1A, Arm1B, and Arm 2

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zucker, Study Chair — Columbia Physicians & Surgeons (P&S) CRS
Locations (9):
- United States (8):
  - Site 5048, USC - Maternal Child Adolescent/Adult Center, Los Angeles, California
  - Site 5112, David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Site 5083, Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Site 4001, Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Site 5040, SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Site 5114, Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Site 5013, Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Site 5128, Baylor College of Medicine/Texas Children's Hospital NICHD CRS, Houston, Texas
- Site 5129, IMPAACT/Gamma Project/UPR Pediatric HIV/AIDS Research CRS, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.